CLINICAL TRIAL: NCT06832982
Title: A Single-arm, Open Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacokinetics, and Preliminary Efficacy of FS-8002 in Patients With Advanced Solid Tumors
Brief Title: Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacokinetics, and Preliminary Efficacy of FS-8002
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pushi Medical Science Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FS-8002-001-CN
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose escalation and dose extension (Experimental): 42patients for dose escalation ,total 6dose group(30 mg、90 mg、270 mg、600 mg、1000 mg、1500 mg），24 patients for dose extension
  Interventions: Drug: FS-8002 injection

INTERVENTIONS:
Drug: FS-8002 injection — Q3W or until the patient develops PD, intolerable toxicity, death, loss of follow-up, voluntary withdrawal, or the end of the study, whichever occurs first

SUMMARY:
this is a single-arm, open phase I clinical trial evaluating the safety, tolerability, pharmacokinetics, pharmacokinetics, and preliminary efficacy of FS-8002 in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced solid tumors confirmed by histology or cytology who have failed or become intolerant to previous standard treatments, or who do not have a standard treatment regimen.GBM patients must be primary GBM and first recurrence after adjuvant radiochemotherapy;
2. According to the evaluation criteria of RECIST V1.1 or RANO 2.0 (GBM only), at least one measurable lesion is required: the selected target lesion has not been treated previously locally, or the selected target lesion is located in the previous local treatment area, but is determined to be disease progression through imaging investigation;
3. The subject has sufficient organ and bone marrow function;

Exclusion Criteria:

1. Patients who have previously received TGF-β inhibitor therapy. previous treatment with bevacizumab or other VEGF or VEGFR-targeted drugs (only for patients with GBM);
2. Have received any experimental drug treatment within 4 weeks prior to the first administration of the investigational drug;
3. Have used any systemic anti-tumor therapy within 4 weeks or 5 half-lives (whichever is shorter) before the first administration of the study drug, including systemic chemotherapy, radiotherapy, immunotherapy, hormone therapy, targeted therapy (small molecule targeted drugs are within 2 weeks before the first administration), systemic immunomodulators (including but not limited to IFN, IL-2 and tumor necrosis factor [TNF]). Received Chinese herbal or proprietary Chinese medicines with anti-tumor effects within 2 weeks before the first administration;For patients with GBM: less than 12 weeks from the end of previous radiotherapy (unless the progressing lesion is located outside the high-dose zone or 80% isodose line irradiation field, or there is pathological evidence), less than 24 days from the last TMZ treatment, or less than 6 weeks from the last carmustine treatment;
4. Have used or are currently using aspirin (≥ 325 mg/day) or other anti-platelet aggregation drugs such as clopidogrel, dipyridamole, ticlopidine, and cilostazole, or full-dose anticoagulants or thrombolytics within 2 weeks prior to the first administration of the study drug;
5. Those who have received major surgical treatment or significant traumatic injury within 4 weeks before the first administration of the study drug, or those who have a history of fistula, gastrointestinal perforation, or tumor invasion of large blood vessels within 6 months before the first administration; or those who have intestinal obstruction during the screening period;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-09-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
MTD | 1.5years
  the maximum tolerated dose(MTD)
RP2D | 1.5years
  the phase II recommended dose(RP2D)
DLT | 1 years
  incidence and serverity of DLT
AE | 2years
  incidence and serverity of adverse events(AE)
SAE | 2years
  incidence and serverity of serious adverse events(SAE)

SECONDARY OUTCOMES:
peak concentration (Cmax) | 1.5years
  the pharmacokinetic parameters of FS-8002: peak concentration (Cmax)
peak time (Tmax) | 1.5years
  the pharmacokinetic parameters of FS-8002: peak time (Tmax)
area under the plasma concentration-time curve (AUC) | 1.5years
  the pharmacokinetic parameters of FS-8002: area under the plasma concentration-time curve (AUC)
T1/2 | 1.5years
  the pharmacokinetic parameters of FS-8002: Terminal half-life
elimination rate constant | 1.5years
  the pharmacokinetic parameters of FS-8002: elimination rate constant
ADA | 1.5years
  Anti-drug antibody
objective response rate (ORR) | 1.5years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate objective response rate (ORR)
disease control rate (DCR) | 1.5years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate disease control rate (DCR)
duration of response (DOR) | 1.5years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate duration of response (DOR)
progression-free survival (PFS) | 1.5years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate progression-free survival (PFS)
overall survival (OS) | 1.5years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate overall survival (OS)

OTHER OUTCOMES:
Cytokines | 1.5years
  Cytokines: interferon gamma (IFN-γ), interleukin (IL) -2, IL-10, IL-12, and IL-15.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer hospital, Fujian, Fuzhou
  - The First Affiliated Hospital of Zhejiang Medical University, Zhejiang, Hangzhou
  - Harbin Medical University Cancer Hospital, Heilongjiang, Harbin
  - Cancer Hospital of Shandong First Medical University(Shandong Cancer Institute,Shandong Cancer Hospital), Shandong, Jinan
  - Meizhou People's Hospital, Guangdong, Meizhou
  - The First Affiliated Hospital of China Medical University, Shenyang, Shenyang
  - Hebei General Hospital, Hebei, Shijiazhuang
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Union Hospital, Tongji Medical College, Hubei, Wuhan
  - Hubei Cancer Hospital, Hubei, Wuhan

IPD SHARING:
Plan to Share IPD: No